CLINICAL TRIAL: NCT04774250
Title: Pharmaceutical Interventions for Noise-Induced Hearing Loss-Acute Exposure Treatment
Brief Title: Noise-Induced Hearing Loss-Acute Exposure Treatment (UA)
Acronym: PINIHL-AET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Texas (Other); Gateway Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PINIHL-AET_UA
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss, Noise-Induced
MeSH Terms: conditions — Hearing Loss, Noise-Induced | interventions — Zonisamide; Capsules; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, and placebo-controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be "masked" or "blinded" in the sense that all the study participants and the study team members will be blinded to the assignment in the study groups. Only the pharmacist who will prepare the drug packets and will seal the envelopes, and the programmer not involved with the study who will produce the random treatment assignments and print the labels will know the order of treatments for any subject. An independent medical professional who is not part of the study team will complete the de-identification of the study drug, and a procedure and documentation log will be in place for quality assurance purposes. The ZNS and placebo capsules will look, taste, and smell the same.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zonisamide (Experimental): For subjects randomized to zonisamide, the package will contain one zonisamide capsule (100 mg PO).
  Interventions: Drug: Zonisamide 100Mg Cap
- Placebo (Placebo Comparator): For the subjects randomized to placebo, the package will contain one placebo capsule that looks, smells, and taste the same as zonisamide capsule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide 100Mg Cap — ZONEGRAN® is commercially available for oral administration as capsules containing 100 mg of Zonisamide.
  Other Names: Zonegran; ZNS
  Arms: Zonisamide
Drug: Placebo — The placebo will contain microcrystalline cellulose which is the predominant filler in the generic capsule.
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of zonisamide (ZNS) for the treatment of noise-induced hearing loss in adults.

DETAILED DESCRIPTION:
This is a randomized, double-blind, and placebo-controlled study is to test whether zonisamide (ZNS) can treat noise-induced hearing loss in police officers on the range following training and certifications sessions. Participants who meet the eligibility requirements will be randomized to receive either ZNS 100 milligrams (mg) or placebo.

Study participants will be recruited from the Akron Police Department, Summit County Police Department, and other local surrounding police departments. Police officers will be offered participation if they are training for firearm certification as part of their standard occupational requirements. These are officers that would be recommended and/or required to complete these trainings/certifications despite this investigation and this investigation will have no influence on audiologic recommendations.

After being informed about the study expectations and potential risks, all individuals providing written informed consent will undergo screening to determine eligibility for study entry.

ELIGIBILITY:
Screening Inclusion Criteria:

* Police officers who are scheduled for firearm training and/or certification on the range.
* At least 18 years of age.
* Air conduction thresholds are to be no worse than 25 dB HL from 0.5 kHz to 3 kHz, no worse than 30 dB HL at 4 kHz, and no worse than 45 dB HL at 6 and 8 kHz prior to shooting range exposure.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Enrollment Inclusion Criteria:

* Observed audiometric TTS ≥ 10 dB HL at 2, 3, 4 and/or 6 kHz
* Observed air-bone gap < 10 dB HL at .5, 1, 2 and 4 kHz, with normal tympanometry

Exclusion Criteria:

* History of known sulfa allergy or hypersensitivity to carbonic anhydrase inhibitors.
* History of moderate-to-severe kidney or liver disease.
* Acute viral, bacterial, fungal or parasitic infection.
* History of seizures.
* Currently pregnant or breast-feeding.
* Any current or history of otologic disorder.
* History of ototoxic drug use.
* Current use of strong/moderate 3A4 inhibitor/inducer and grapefruit juice.
* For secondary outcomes, exclusion criteria is as follows:

  1. DPOAE data will be used as a secondary outcome measure of TTS, and participants will be excluded if their DPOAE is absent at more than 3/7 frequencies. Criteria for a present response is any response that is > 5 dB SPL above the noise floor and replicable within ±5 dB SPL.
  2. ECochG: Participants will be excluded if the ECochG/ABR wave I response is absent.
  3. WIN test: Participants with WIN scores greater than moderate difficulty or 14.9 dB SNR will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Buchman, MD, FACS, Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Akron, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (0) | 37 (6) | 39 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Officers With Permanent Threshold Shift (PTS)
Description: The proportion of PTS-positive subjects defined as the ratio of PTS-positive subjects to total number of subjects within each study arm/group. Subjects defined as PTS-positive will demonstrate an increase in threshold that is ≥10 dB HL at any frequency from 2-6 kHz post-shooting as compared to baseline audiogram.
Time Frame: 30 days (+/- 3 days) after training
Population: The study was prematurely terminated. Due to the very low number of subjects in each study group there was no statistical analysis performed; no statistical test, p-value, or parameter estimation can be reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 1 | 2
Participants
  PTS-positive participants | 0 | 1
  PTS-negative participants | 1 | 1

2. Secondary Outcome: Distortion Product Otoacoustic Emissions (DPOAE)
Description: DPOAE amplitudes are measured to determine threshold shifts. A change is noted in DPOAE amplitude at any frequency that is significantly greater than the stability of each measurement (i.e., 95% confidence interval of each measurement do not overlap).
Time Frame: baseline (before shooting), 30 days (+/-3 days) after training
Population: Each participant's left and right ears were analyzed for threshold shifts at 30 days (+/- 3 days) after training.
Measure: Count of Units; unit: ears
Units Other Than Participants: ears
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 1 | 2
Number analyzed (ears) | 2 | 4
ears
  No Shift | 1 | 0
  Shift | 1 | 3
  Excluded | 0 | 1

3. Secondary Outcome: Ultra-high Frequency Audiometry
Description: Number of participants that experience a change in ultra-high frequencies greater than 5 dB; to measure for both temporary and permanent high frequency audiometric changes. A significant change is defined for any frequency that is greater than 5 dB HL from baseline thresholds.
Time Frame: baseline (before shooting), within 5-10 minutes after shooting and 30 days (+/-3 days) after training
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 1 | 2
Participants
  Experienced a change in ultra-high frequencies greater than 5 dB | 1 | 2
  Did not experience a change in ultra-high frequencies greater than 5 dB | 0 | 0

4. Secondary Outcome: Electrocochleography (ECochG) AP Amplitude
Description: To measure for changes in ECochG AP amplitude between baseline (before training) visit and 30-days after training visits.
Time Frame: baseline (before shooting) and 30 days (+/-3 days) after training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 1 | 2
millivolts (mV) | 0.035 (0) | 0.1025 (0.159)

5. Secondary Outcome: Change in Words In Noise (WIN) Test Signal-to-Noise Ratio Threshold
Description: The WIN test battery consists of 35 words that are presented in a background noise (speech babble) with varying degrees of signal-to-noise ratios (SNR) from 24 dB HL to 0 dB HL. The WIN score will be repeated three times in order to assess test-retest reliability. The total number of words correctly identified will be used to calculate a dB HL S/N threshold by the Spearman-Karber equation at the mean of 50% correct points. Reported information is the change in score between baseline testing and testing 30 days after training.
  This measure assesses the change in signal-to-noise ratio (SNR) threshold, reported in decibels SNR (dB SNR), at which a participant correctly identifies 50% of the words presented in background noise.
Time Frame: baseline (before shooting) and 30 days (+/-3 days) after training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB SNR
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 1 | 2
dB SNR | -0.267 (0) | 1.933 (0.660)

6. Secondary Outcome: Electrocochleography (ECochG) Latency
Description: To measure for changes in ECochG latency between baseline (before training) visit and 30-days after training visits.
Time Frame: baseline (before shooting) and 30 days (+/-3 days) after training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 1 | 2
milliseconds (ms) | 0.105 (0) | -0.053 (0.046)

7. Secondary Outcome: Electrocochleography (ECochG) Width
Description: To measure for changes in ECochG width between baseline (before training) visit and 30-days after training visits.
Time Frame: baseline (before shooting) and 30 days (+/-3 days) after training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 1 | 2
milliseconds (ms) | 0.295 (0) | 0.030 (0.028)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Documentation of adverse events at all follow-up visits (5-30 minutes post, within 24 hours, and at 30 day visit; follow-up visit 3, 4, and 5).
  Adverse events were tracked post dose within 30 minutes, 24 hours, and at 30 days. All adverse events were recorded on an Adverse Events tracking case report form (CRF). Adverse events related to study medication only were tracked.
Arm/Group | Zonisamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to the low number of eligible subjects (3 subjects); therefore, statistical analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT04774250/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT04774250/SAP_001.pdf